CLINICAL TRIAL: NCT01763814
Title: A Randomized, Single Blind Study of the Efficacy and Safety of Three Different Approaches for Ultrasound Guided Femoral Nerve Block for Patients Undergoing Total Knee Arthroplasty
Brief Title: Three Different Approaches for Ultrasound Guided Femoral Nerve Block for Patients Undergoing Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chicago Anesthesia Pain Specialists (Other)
Responsible Party: Principal Investigator, Antony Tharian, MD, Chicago Anesthesia Pain Specialists
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Advocate-IRB-5235
Record Dates: First submitted 2013-01-02; First posted 2013-01-09 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Knee Arthroplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Single shot femoral nerve block (Active Comparator): A ultrasound probe will be used to identify the nerve, and correct needle placement.
  Interventions: Procedure: Femoral nerve block
- Femoral nerve block non stimulating catheter (Active Comparator): A ultrasound probe will be used to identify the nerve, and correct needle placement. The catheter will be placed with the nerve stimulator powered off.
  Interventions: Procedure: Femoral nerve block; Procedure: Femoral nerve block non stimulating catheter
- Femoral nerve block stimulating catheter (Active Comparator): A ultrasound probe will be used to identify the nerve, and correct needle placement. The catheter will be placed with the nerve stimulator powered on.
  Interventions: Procedure: Femoral nerve block; Procedure: Femoral nerve block stimulating catheter

INTERVENTIONS:
Procedure: Femoral nerve block — A visible or palpable cephalad movement of the patella will confirm needle placement.
Procedure: Femoral nerve block non stimulating catheter — A visible or palpable cephalad movement of the patella will confirm needle placement. The catheter will be placed with the nerve stimulator powered off.
  Arms: Femoral nerve block non stimulating catheter
Procedure: Femoral nerve block stimulating catheter — A visible or palpable cephalad movement of the patella will confirm needle placement. The catheter will be placed with the nerve stimulator powered on.
  Arms: Femoral nerve block stimulating catheter

SUMMARY:
Patients scheduled to have a surgery for Total Knee Arthroplasty will be assigned to one of three groups, each group will use a different approach using the ultrasound to guide the femoral nerve block as part of their treatment for controlling pain post-operatively.

DETAILED DESCRIPTION:
This will be a prospective, single-blinded, randomized study. The patients will be randomly assigned to one of three groups:

Group I - single shot femoral nerve block Group II - continuous femoral nerve block - non stimulating catheter Group III - continuous femoral nerve block - stimulating catheter

ELIGIBILITY:
Inclusion Criteria:

* 18- 90 years old
* Scheduled for total knee arthroplasty

Exclusion Criteria:

* Redo surgery on the same knee
* BMI ≥45
* Radicular pain in the same leg
* Allergy to local anesthetics
* Opioid habituation
* Pregnancy
* Contraindication to regional block
* Inability to communicate with hospital staff or investigators.
* Neuropathy of any etiology in the surgical extremity.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-12; Primary Completion 2018-02 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change in the Numeric Rating Pain Score | Postoperative
  At the conclusion of the surgery time 0, at 15, 30, and 45 minutes, at 1, 12, 24, 48 hours, and day 3, 7, 14, and 30 after the surgery.

SECONDARY OUTCOMES:
Change in the ability to move the knee | Postoperative
  At the conclusion of the surgery time 0, at 15, 30, and 45 minutes, at 1, 12, 24, 48 hours, and day 3, 7, 14, and 30 after the surgery.
Change in Supplemental pain medications | Postoperative
  At the conclusion of the surgery time 0, at 15, 30, and 45 minutes, at 1, 12, 24, 48 hours, and day 3, 7, 14, and 30 after the surgery.

OTHER OUTCOMES:
Change in the overall satisfaction | Postoperative
  At the conclusion of the surgery time 0, at 15, 30, and 45 minutes, at 1, 12, 24, 48 hours, and day 3, 7, 14, and 30 after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Antony Tharian, M.D., Principal Investigator — Chicago Anesthesia Pain Specialists
Locations (1):
- Chicago Anesthesia Pain Specialists, Chicago, Illinois, United States